CLINICAL TRIAL: NCT01710254
Title: Detection of Coronary Artery Disease in Patients With Atrial Fibrillation Using Regadenoson Stress MRI
Brief Title: Regadenoson Stress-MRI to Identify Coronary Artery Disease in Atrial Fibrillation Patients
Acronym: RECAD-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brent Wilson, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REGA-12F08
Record Dates: First submitted 2012-10-02; First posted 2012-10-19 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease
Keywords: MRI; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease | interventions — regadenoson; gadobenic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regadenoson MRI (Experimental): Participants with AF receiving regadenoson stress MRI, using Gadobenate dimeglumine
  Interventions: Drug: Regadenoson MRI; Drug: Gadobenate dimeglumine

INTERVENTIONS:
Drug: Regadenoson MRI — AF patients will be provided with a regadenoson stress MRI to see if coronary artery disease can be detected with more sensitivity /specificity.
  Other Names: Lexiscan
Drug: Gadobenate dimeglumine — Resting perfusion with Multihance Gd-BOPTA contrast agent will be performed first, then a regadenoson injection will be given and MR imaging performed with a Gd-BOPTA contrast agent bolus 60-100 seconds later.
  Other Names: Gd-BOPTA; Multihance

SUMMARY:
Atrial fibrillation (AF) is growing into an epidemic affecting 1 in 4 adults. There is a need for research to elucidate the prevalence of ischemic cardiomyopathy in patients diagnosed with AF. The objective of this study is to demonstrate the utility of MRI in assessment of coronary artery disease. The specific objective is to demonstrate sensitivity/specificity comparable to that reported in meta-analyses of non-AF patients and adenosine (90% /80%) in an AF population using the time-efficient vasodilator regadenoson that requires only a single intravenous (IV).

DETAILED DESCRIPTION:
Scientific Background/Rationale:

Atrial fibrillation (AF) is a large and growing healthcare problem worldwide. Over 7 million people in the U.S. and Europe currently suffer from atrial fibrillation, and this number is expected to double before 2050. The lifetime risk of AF is high: ~24% at age 40, and this risk remains fairly constant at older ages, with 22% lifetime risk at age 80 [1]. AF significantly increases the risk of stroke and mortality, and can greatly limit quality of life. Little research has been done on AF and ischemic cardiomyopathy, though it is a relatively common co-morbidity. CT found increased prevalence (41% vs 27%) of coronary artery disease (CAD) in patients with AF compared to patients with similar pre-test risk but no AF [2]. AF patients with a positive SPECT scan for CAD have a worse prognosis for cardiac events than patients with positive SPECT but without AF [3]. It was recently reported that in a study of 253 AF patients, that AF patients with positive SPECT studies had a very high number of false positives - only 15% of patients had significant CAD by angiography (compared to 67% in the control group) [4, 5]. Just over half of the patients were in sinus rhythm at SPECT, but since similar numbers of positives were seen in each half, the authors did not feel that imaging during AF was the cause of the poor specificity.

Use of MRI for assessment of CAD is a growing area that entails no radiation exposure to the patient. Advances in MRI have made it possible to accurately detect CAD, either as well or better than SPECT in unselected populations [6, 7]. However, adoption of MRI myocardial perfusion scans has been limited in part due to the challenges associated with the use of adenosine. Adenosine requires starting a second IV, and to use either a special expensive MRI-compatible infusion pump to deliver the drug, or long lengths of tubing to run to a pump outside the scanner room. Neither solution is ideal, and regadenoson would not require any such pumps or the starting of a second IV. Here the investigators propose to determine the sensitivity/specificity for dynamic contrast-enhanced myocardial perfusion MRI with the vasodilator regadenoson in a subpopulation of patients - those with atrial fibrillation.

The investigators have a great deal of experience with stress and rest myocardial perfusion MRI. In a preliminary study imaging three patients with AF that then went to X-ray angiography (cath), two of the three subjects had significant stenoses by cath, and one did not. This agreed with the regadenoson stress perfusion MRI findings. These MRI acquisitions were performed on a Siemens Verio MRI scanner. The Verio operates at twice the magnetic field strength (3 Tesla, or 3T) of most MRI scanners, which operate at 1.5T. The higher magnetic field offers images with significantly less noise (almost twice the signal-to-noise ratio).

Objective: To demonstrate sensitivity/specificity comparable to that reported in meta-analyses of non-AF patients and adenosine (90%/80% [6, 7]), in an atrial fibrillation population while using the time-efficient vasodilator regadenoson that requires only a single IV.

Study Design: This will be a prospective, open-label, comparative trial using MRI. Non-invasive MRI measurements of resting flow and flow at regadenoson stress will be obtained in each subject during a one hour MRI exam using our advanced MRI acquisition techniques. Sensitivity/specificity of regadenoson stress MRI will be determined using x-ray angiography as the standard. X-ray angiography will be done as standard-of-care, and is not an intervention of this clinical trial.

Study Procedure: Each subject will undergo a single MRI scanning session. Caffeine will be stopped 12 hours prior to the procedure. One IV will be started and subjects positioned in the scanner. Resting perfusion with Multihance Gd-BOPTA contrast agent will be performed first. The perfusion acquisition acquires 3-6 short axis slices each heartbeat and lasts for one minute. Then a standard regadenoson injection of 400ug/5cc will be given and MR imaging performed with a Gd-BOPTA contrast agent bolus 60-100 seconds later [9] [10].

ELIGIBILITY:
Inclusion Criteria:

Patients with confirmed persistent or paroxysmal AF and suspected coronary artery disease who will undergo catheterization X-ray angiography

Exclusion Criteria:

1. Critically ill patients, patients on ventilators patients with hypotension, asthmatics, and other patients whose medical care or safety may be compromised from undergoing an MRI examination will be excluded.
2. Patients with claustrophobia will also be excluded since MRI is conducted in a closed environment.
3. Patients with contraindications to MRI (pacemaker, metal implants).
4. Pregnant subjects (or women who may become pregnant), minors, and prisoners will be excluded from this study.
5. Subjects are over 60 or have any suspicion of abnormal kidney function (a blood test to determine Glomerular filtration rate (GFR) will be performed prior to imaging. Subjects with GFR<30 will be excluded from the study. This is standard practice for clinical scans in Radiology due to the extremely small but not negligible relationship between gadolinium contrast agent and nephrogenic systemic fibrosis in patients with severely impaired renal function.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Wilson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Background] Nucifora G, Schuijf JD, Tops LF, van Werkhoven JM, Kajander S, Jukema JW, Schreur JH, Heijenbrok MW, Trines SA, Gaemperli O, Turta O, Kaufmann PA, Knuuti J, Schalij MJ, Bax JJ. Prevalence of coronary artery disease assessed by multislice computed tomography coronary angiography in patients with paroxysmal or persistent atrial fibrillation. Circ Cardiovasc Imaging. 2009 Mar;2(2):100-6. doi: 10.1161/CIRCIMAGING.108.795328. Epub 2009 Jan 26. PMID 19808575
- [Background] Abidov A, Hachamovitch R, Rozanski A, Hayes SW, Santos MM, Sciammarella MG, Cohen I, Gerlach J, Friedman JD, Germano G, Berman DS. Prognostic implications of atrial fibrillation in patients undergoing myocardial perfusion single-photon emission computed tomography. J Am Coll Cardiol. 2004 Sep 1;44(5):1062-70. doi: 10.1016/j.jacc.2004.05.076. PMID 15337220
- [Background] Smit MD, Tio RA, Slart RH, Zijlstra F, Van Gelder IC. Myocardial perfusion imaging does not adequately assess the risk of coronary artery disease in patients with atrial fibrillation. Europace. 2010 May;12(5):643-8. doi: 10.1093/europace/eup404. Epub 2009 Dec 17. PMID 20022875
- [Background] Nandalur KR, Dwamena BA, Choudhri AF, Nandalur MR, Carlos RC. Diagnostic performance of stress cardiac magnetic resonance imaging in the detection of coronary artery disease: a meta-analysis. J Am Coll Cardiol. 2007 Oct 2;50(14):1343-53. doi: 10.1016/j.jacc.2007.06.030. Epub 2007 Sep 17. PMID 17903634
- [Background] Hamon M, Fau G, Nee G, Ehtisham J, Morello R, Hamon M. Meta-analysis of the diagnostic performance of stress perfusion cardiovascular magnetic resonance for detection of coronary artery disease. J Cardiovasc Magn Reson. 2010 May 19;12(1):29. doi: 10.1186/1532-429X-12-29. PMID 20482819
- [Background] Ablitt NA, Gao J, Keegan J, Stegger L, Firmin DN, Yang GZ. Predictive cardiac motion modeling and correction with partial least squares regression. IEEE Trans Med Imaging. 2004 Oct;23(10):1315-24. doi: 10.1109/TMI.2004.834622. PMID 15493698
- [Background] S. E. Litwin, J. Fluckiger, L. Chen, T. H. Kim, N. Pack, B. Matthews, C. McGann, R. Jiji, et al. Does fixed-dose regadenoson induce comparable myocarial perfusion reserve in patients of widely varying body size? A quantitative MRI study. American Heart Association, chicago, 2010.
- [Background] O. J. Booker, P. Bandettini, P. Kellman, J. Wilson, S. Leung, S. Vasu, S. Shanbhag, J. Henry, et al. Time resolved measure of coronary sinus flow following regadenoson administration. Journal of cardiovascular magnetic resonance, 13(1): O74, 2011.
- [Background] Harper R, Reeves B. Reporting of precision of estimates for diagnostic accuracy: a review. BMJ. 1999 May 15;318(7194):1322-3. doi: 10.1136/bmj.318.7194.1322. No abstract available. PMID 10323817
- [Derived] Bieging ET, Haider I, Adluru G, Chang L, Suksaranjit P, Likhite D, Shaaban A, Jensen L, Wilson BD, McGann CJ, DiBella E. Rapid rest/stress regadenoson ungated perfusion CMR for detection of coronary artery disease in patients with atrial fibrillation. Int J Cardiovasc Imaging. 2017 Nov;33(11):1781-1788. doi: 10.1007/s10554-017-1168-1. Epub 2017 May 20. PMID 28528431

RESULTS

PARTICIPANT FLOW:
Groups:
- Regadenoson MRI: Participants with atrial fibrillation receiving regadenoson stress MRI
Period: Overall Study
Arm/Group | Regadenoson MRI
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regadenoson MRI
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Regadenoson Stress-MRI for Detection of Coronary Artery Disease (CAD)
Description: Determination of sensitivity of Regadenoson stress-MRI in the detection of CAD, using x-ray angiography as the standard. Perfusion images interpreted by three blinded readers as normal or abnormal; majority results of the three blinded readers are reported.
Time Frame: one MRI, up to 1 hour
Population: Results for 4 subjects are unevaluable due to delays in blinded reading of MRI scans and non-comparable due to personnel turnover in blinded MRI readers
Measure: Number (95% Confidence Interval); unit: Percentage of true positive cases
Arm/Group | Regadenoson MRI
Number analyzed (Participants) | 26
Percentage of true positive cases | 80 [30 to 99]

2. Primary Outcome: Specificity of Regadenoson Stress-MRI for Detection of Coronary Artery Disease (CAD)
Description: Determination of specificity of Regadenoson stress-MRI in the detection of CAD, using x-ray angiography as the standard. Perfusion images interpreted by three blinded readers as normal or abnormal; majority results of the three blinded readers are reported.
Time Frame: one MRI, up to 1 hour
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of true negative cases
Arm/Group | Regadenoson MRI
Number analyzed (Participants) | 26
Percentage of true negative cases | 100 [81 to 100]

3. Secondary Outcome: Accuracy of Regadenoson Stress-MRI for Detection of Coronary Artery Disease (CAD)
Description: Determination of accuracy of Regadenoson stress-MRI in the detection of CAD, using x-ray angiography as the standard. Accuracy is the percentage of correctly classified subjects (true positive + true negative) among all subjects (true positive + true negative + false positive + false negative). Perfusion images interpreted by three blinded readers as normal or abnormal; majority results of the three blinded readers are reported.
Time Frame: one MRI, up to 1 hour
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of correct total cases
Arm/Group | Regadenoson MRI
Number analyzed (Participants) | 26
Percentage of correct total cases | 96 [78 to 100]

ADVERSE EVENTS:
Time Frame: Subjects monitored for safety events during the entire magnetic resonance imaging session; up to 1 hour
Arm/Group | Regadenoson MRI
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 15/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regadenoson MRI (N=30)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Headache (Nervous system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No